CLINICAL TRIAL: NCT04891432
Title: Comparison of Surgical Outcomes Between Pre Sympathetic Plexus and Post Sympathetic Plexus Approach
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chi Heon Kim, Professor, Seoul National University Hospital
Other Study IDs: 2101-142-1191
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Fusion of Spine; Sympathetic Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Procedure: Lateral lumbar interbody fusion — oblique lumbar interbody fusion or direct lateral interbody fusion
  Other Names: front versus back sympathetic chain approach

SUMMARY:
There would be no difference in the risk of sympathetic plexus damage between the pre sympathetic plexus approach and the post sympathetic plexus approach.

DETAILED DESCRIPTION:
Compare the incidence of sympathetic chain injury between front and back of sympathetic approach in oblique lumbar interbody fusion

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar degenerative disease needs a lateral lumbar interbody fusion of 1-2 segments between L2 to S1.

Exclusion Criteria:

* Patients who had previously had lumbar surgery
* Patients with muscle weakness of motor grade III or lower
* Patients with neuropsychiatric diseases such as depression
* Patients with musculoskeletal disease, inflammatory musculoskeletal disease, or infection
* Patients with cancerous disease
* Patients who do not want to participate in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lumbar degenerative disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of sympathetic plexus injury | Postoperative day one
  The number of patiensts with sympathetic symptom such as edema of the lower extremity, change of skin temperature, pain, or paresthesia without other medical conditions

SECONDARY OUTCOMES:
Other complications | Postoperative 6 month
  the number of patients with any other complication such as Injury of vascular structure, ureter, peritoneum, or bowel.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No